CLINICAL TRIAL: NCT00474682
Title: Relative Bioavailability of Ferric Pyrophosphate From an Apple Juice Drink
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quadram Institute Bioscience (Other)
Collaborators: The Coca-Cola Company (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: IFR04/2006
Record Dates: First submitted 2007-05-16; First posted 2007-05-17 (Estimated); Last update posted 2008-12-03 (Estimated); Status verified 2007-05

CONDITIONS: Iron Deficiency
Keywords: ferric pyrophosphate, iron bioavailability, fortification,
MeSH Terms: conditions — Iron Deficiencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Micronized dispersible ferric pyrophosphate

SUMMARY:
The aim of this study is to find out how well iron is absorbed when a newly developed form of ferric pyrophosphate is added to a commercial apple juice drink.

DETAILED DESCRIPTION:
Micronized dispersible ferric pyrophosphate (MDFP) is an iron compound that has been reported to be highly bioavailable and likely to cause few sensory problems when added to food. It is therefore a potentially effective iron additive for the food industry and is particularly formulated for adding to liquids. A randomized cross-over trial will be undertaken to compare the absorption of iron added to a commercial apple juice drink as MDFP with iron added as ferrous sulphate. The null hypothesis is that absorption of iron added as MDFP is not different to absorption from iron added as ferrous sulphate.

The study population will consist of 16 women (age 18-65) with iron stores at the lower end of the normal range. This group will efficiently absorb bioavailable iron and will be sensitive to differences in bioavailability between different forms of iron. Test drinks containing added iron, labelled with stable isotopes of iron (Fe-57 or Fe-58), will be consumed on two consecutive days. Iron absorption from the drinks will be determined using the erythrocyte incorporation technique. A baseline blood sample will be taken prior to consuming the test drinks and then a second blood sample will be taken 14 days after the last test drink. Iron absorption will be calculated from the isotopic enrichment of the final blood sample, assuming that 80% of absorbed iron is incorporated into red blood cells. The order in which the volunteers will be given the MDFP or ferrous sulphate will be randomised.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Age >18 and <65
* BMI >18.5 and <35
* Serum ferritin value of =12μg/L and =50μg/L

Exclusion Criteria:

* Men
* Age < 18 or >65
* BMI <18.5 or >35
* Serum ferritin value of <12μg/L or >50μg/L
* Volunteers will be excluded if they are found to have depressed or elevated blood pressure measurements (<90/50 or<95/50 if symptomatic or >160/100)
* Diagnosed with a long-term illness requiring active treatment, e.g. diabetes, cancer, cardiovascular disease
* Gastrointestinal disease (excluding hiatus hernia unless symptomatic)
* Regular prescribed medication that may interfere with iron metabolism
* Regular use of antacids and laxatives (at least once a week)
* Women who are pregnant or less than 12 months since giving birth
* Women breast feeding
* Vitamin supplements with or without minerals if taken more than once a week, and unwillingness to discontinue occasional use for the duration of study
* Unwillingness to discontinue use of herbal supplements for the duration of study
* Use of antibiotics within four weeks prior to study start
* Parallel participation in another study which involves dietary interventions or sampling of blood that may increase the volume taken above 500ml in a 4-month period.
* Asthma requiring treatment within the last two years
* Results of clinical screening which indicate, or are judged by the HNU Medical advisor to be indicative of a health problem which could compromise the well-being of the volunteer if they participated or which would affect the study data.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)

PRIMARY OUTCOMES:
Relative bioavailability of Micronized dispersible ferric pyrophosphate added to apple juice | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Susan J Fairweather-Tait, Principal Investigator — University of East Anglia
Locations (1):
- Institute of Food Research, Norwich, Norfolk, United Kingdom